CLINICAL TRIAL: NCT04131933
Title: A Multi-centre, Prospective, Observational Study Evaluating Whether Integration of Prognostic and Predictive Algorithms Into Routine Clinical Practice Effect Whether Oncologists Order Multigene Assays in Patients With Early Stage Breast Cancer
Brief Title: Evaluating Whether Integration of Prognostic and Predictive Algorithms Into Routine Clinical Practice Effect Whether Oncologists Order Multigene Assays in Patients With Early Stage Breast Cancer
Acronym: REaCT-Algorith
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: REaCT-Algorithm
Record Dates: First submitted 2019-10-01; First posted 2019-10-18 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Predict 2.1; Oncotype DX
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A broad range of prognostic and predictive tools are available for patients with newly diagnosed early stage breast cancer. These range from free and publicly available mathematical algorithms, through to expensive genomic tests. It is not known how the use of these different scores affects physician decision making with respect to ordering genomic tests, nor how well these algorithms predict for the results of Oncotype DX ® in the real-world setting. This pragmatic study will help to answer these questions.

DETAILED DESCRIPTION:
A broad range of prognostic and predictive tools are available for patients with newly diagnosed early stage hormone receptor positive, Her2 negative breast cancer. These range from free and publicly available mathematical algorithms (e.g. NHS Predict, Magee formulae, Gage and Tennessee equations) that incorporate standard pathology results, through to expensive genomic tests (e.g. Oncotype DX ® and Endopredict ®). It is not known how the use of these different scores affects physician decision making with respect to ordering genomic tests, nor how well these algorithms predict for the results of Oncotype DX ® in the real-world setting. This pragmatic study will help to answer these questions.

In summary: Month 1 to 3: pathology and chemotherapy data is collected, no physician questionnaires given. Month 4 to 6: pathology and chemotherapy data collected, plus physician questionnaire administered. Intervention teaching after 6 months of study activation. Month 7 to 9: pathology and chemotherapy data collected, PREDICT 2.1 tool used, no physician questionnaire given. Month 10 to 12: pathology and chemotherapy data collected, PREDICT 2.1 tool used, plus physician questionnaire administered.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary breast cancer
* No prior chemotherapy
* Eligible for Oncotype DX ® testing as per current Ontario funding criteria including: ER positive, PR positive or negative, HER2 negative, lymph node status negative or micro-invasive disease, tumor >1 cm in size (or if equal or <1 cm, must be grade 2/3 or have lymph node micrometastasis).

Exclusion Criteria:

* Neoadjuvant treatment including window of opportunity trials
* Recurrent breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are eligible for Oncotype DX ® testing under current funding parameters with complete pathology reports for newly diagnosed early stage breast cancer will be eligible for this prospective trial.
Sampling Method: Non-Probability Sample
Enrollment: 602 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arif Awan, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (6):
- Canada (6):
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Grand River Hospital, Kitchener, Ontario
  - Markham Stouffville Hospital, Markham, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Windsor Regional Hospital, Windsor, Ontario

REFERENCES:
- [Background] Robertson SJ, Ibrahim MFK, Stober C, Hilton J, Kos Z, Mazzarello S, Ramsay T, Fergusson D, Vandermeer L, Mallick R, Arnaout A, Dent SF, Segal R, Sehdev S, Gertler S, Hutton B, Clemons M. Does integration of Magee equations into routine clinical practice affect whether oncologists order the Oncotype DX test? A prospective randomized trial. J Eval Clin Pract. 2019 Apr;25(2):196-204. doi: 10.1111/jep.13094. Epub 2019 Jan 23. PMID 30672056
- [Background] de Lima MAG, Clemons M, Van Katwyk S, Stober C, Robertson SJ, Vandermeer L, Fergusson D, Thavorn K. Cost analysis of using Magee scores as a surrogate of Oncotype DX for adjuvant treatment decisions in women with early breast cancer. J Eval Clin Pract. 2020 Jun;26(3):889-892. doi: 10.1111/jep.13223. Epub 2019 Jul 9. PMID 31287198
- [Background] Robertson SJ, Pond GR, Hilton J, Petkiewicz SL, Ayroud Y, Kos Z, Gravel DH, Stober C, Vandermeer L, Arnaout A, Clemons M. Selecting Patients for Oncotype DX Testing Using Standard Clinicopathologic Information. Clin Breast Cancer. 2020 Feb;20(1):61-67. doi: 10.1016/j.clbc.2019.07.006. Epub 2019 Aug 22. PMID 31551182
- [Result] Awan AA, Saunders D, Pond G, Hamm C, Califaretti N, Mates M, Kumar V, Ibrahim MFK, Beltran-Bless AA, Vandermeer L, Hilton J, Clemons M. Does Pre-Emptive Availability of PREDICT 2.1 Results Change Ordering Practices for Oncotype DX? A Multi-Center Prospective Cohort Study. Curr Oncol. 2024 Feb 27;31(3):1278-1290. doi: 10.3390/curroncol31030096. PMID 38534929
- See also: The Rethinking Clinical Trials (REaCT) website — https://react.ohri.ca/

RESULTS

PARTICIPANT FLOW:
Groups:
- Period 1: Patients who were seen with clinical and pathological features in Months 0-3
- Period 2: Patients who were seen with clinical and pathological features in Months 4-6
- Period 3: Patients who were seen with clinical and pathological features in Months 7-9
- Period 4: Patients who were seen with clinical and pathological features in Months 10-12
Period: Overall Study
Arm/Group | Period 1 | Period 2 | Period 3 | Period 4
Started | 198 | 123 | 125 | 156
Completed | 198 | 123 | 125 | 156
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Period 1 | Period 2 | Period 3 | Period 4 | Total
Number analyzed (Participants) | 198 | 123 | 125 | 156 | 602
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (12.6) | 64.5 (11.7) | 64.6 (11.2) | 62.3 (11.2) | 63.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 122 | 124 | 153 | 596
  Male | 1 | 1 | 1 | 3 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Oncotype DX Testing Ordered
Description: To assess whether providing individual patient prognostic and predictive scores from PREDICT 2.1 affects the rate of subsequent requests for Oncotype DX ® testing.
  This is measured as the number of participants with Oncotype DX ® testing ordered.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1 | Period 2 | Period 3 | Period 4
Number analyzed (Participants) | 198 | 123 | 125 | 156
Participants | 92 | 62 | 50 | 74
Statistical Analysis 1: Comparison: Period 1 vs Period 2 vs Period 3 vs Period 4; Pre-Intervention (Period 1 and Period 2) vs Post-Intervention (Period 3 and Period 4); Test type: Superiority — It was hypothesized that there would be a 50% reduction in Oncotype DX assay requests following the intervention; p = 0.37, Fisher Exact; Fisher's exact test to compare number of patients with Oncotype DX ordered at 0-6 months (pre-intervention) vs 7-12 months (post-intervention)

2. Secondary Outcome: Time From Resection to Treatment
Description: To assess whether routine availability of PREDICT 2.1 affects adjuvant treatment (chemotherapy, radiation therapy and endocrine therapy). This will be done by identifying the time to starting chemotherapy, endocrine therapy or radiation therapy.
Time Frame: 12 Months
Population: The overall number of participants analyzed are the number of participants in each period. Each row in the outcome measure data table has a different number of participants analyzed per period because not every participant received each treatment type (chemotherapy, radiation, endocrine therapy).
Measure: Median (Full Range); unit: months
Arm/Group | Period 1 | Period 2 | Period 3 | Period 4
Number analyzed (Participants) | 198 | 123 | 125 | 156
months
  Resection to chemotherapy: number analyzed (Participants) | 22 | 10 | 14 | 23
  Resection to chemotherapy | 1.9 [1.0 to 3.0] | 1.8 [0.2 to 2.5] | 1.8 [1.3 to 2.4] | 1.9 [0.7 to 3.2]
  Resection to radiation: number analyzed (Participants) | 112 | 88 | 90 | 110
  Resection to radiation | 2.4 [1.0 to 7.9] | 2.2 [1.0 to 8.1] | 2.1 [1.0 to 6.2] | 2.3 [0.9 to 9.1]
  Resection to endocrine therapy: number analyzed (Participants) | 169 | 104 | 110 | 130
  Resection to endocrine therapy | 1.8 [0.0 to 8.2] | 1.9 [0.5 to 7.1] | 2.3 [0.6 to 7.6] | 2.2 [0.5 to 9.8]

3. Secondary Outcome: Oncotype DX ® Cost
Description: Prognostic risk scores, including Magee formulae, Gage and Tennessee equations will be calculated using patient and tumour characteristics. These scores will be compared with Oncotype DX ® scores when performed. These will be used to determine Oncotype DX ® cost and total health system costs and subsequent health care utilization.
Time Frame: 12 Months
Reporting Status: Not Posted, anticipated posting 2027-12

4. Secondary Outcome: Physician Survey
Description: A physician survey will be used to assess physician comfort when making systemic therapy decisions.It will determine whether the routine availability of PREDICT 2.1 score in the clinic enhanced their comfort with systemic therapy decision-making.
Time Frame: Period 2 (Months 4-6) and Period 4 (Months 10-12)
Population: Survey was only administered in Period 2 and Period 4. The number analyzed for each row differs from the overall number of participants analyzed because some surveys may have been incomplete and some items left unanswered.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1 | Period 2 | Period 3 | Period 4
Number analyzed (Participants) | 0 | 123 | 0 | 156
Participants
  PREDICT results make me more confident in my recommendation: number analyzed (Participants) | 0 | 62 | 0 | 149
  PREDICT results make me more confident in my recommendation: Strongly Disagree | 0 | 1 | 0 | 3
  PREDICT results make me more confident in my recommendation: Disagree | 0 | 8 | 0 | 12
  PREDICT results make me more confident in my recommendation: Neither Agree nor Disagree | 0 | 10 | 0 | 32
  PREDICT results make me more confident in my recommendation: Agree | 0 | 31 | 0 | 71
  PREDICT results make me more confident in my recommendation: Strongly Agree | 0 | 12 | 0 | 31
  PREDICT tool influenced my treatment decision: number analyzed (Participants) | 0 | 72 | 0 | 153
  PREDICT tool influenced my treatment decision: Strongly Disagree | 0 | 3 | 0 | 7
  PREDICT tool influenced my treatment decision: Disagree | 0 | 11 | 0 | 21
  PREDICT tool influenced my treatment decision: Neither Agree nor Disagree | 0 | 17 | 0 | 47
  PREDICT tool influenced my treatment decision: Agree | 0 | 32 | 0 | 56
  PREDICT tool influenced my treatment decision: Strongly Agree | 0 | 9 | 0 | 22
  I would use PREDICT tool again: number analyzed (Participants) | 0 | 73 | 0 | 153
  I would use PREDICT tool again: Strongly Disagree | 0 | 1 | 0 | 1
  I would use PREDICT tool again: Disagree | 0 | 1 | 0 | 5
  I would use PREDICT tool again: Neither Agree nor Disagree | 0 | 3 | 0 | 19
  I would use PREDICT tool again: Agree | 0 | 41 | 0 | 68
  I would use PREDICT tool again: Strongly Agree | 0 | 27 | 0 | 60

ADVERSE EVENTS:
Time Frame: Adverse events were not collected.
Description: Adverse events were not collected.
Arm/Group | Period 1 | Period 2 | Period 3 | Period 4
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/33/NCT04131933/Prot_SAP_000.pdf